CLINICAL TRIAL: NCT00264173
Title: A Twelve-Week, Open, Randomized Trial Comparing Valproate to Lithium in Bipolar I Patients Suffering From a Manic Episode
Brief Title: VALID : VAlproate Versus LIthium in Bipolar Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R_8740
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

INTERVENTIONS:
Drug: Valproate sodium

SUMMARY:
Primary Objective :

* To compare the efficacy of valproate to lithium in Bipolar I patients suffering from a manic or a mixed episode according to DSM IV TR (APA 2000) [Diagnostic and Statistical Manual of Mental Disorders (DSM) fourth edition (IV)Text Revision (TR)] and over a periode of 3 weeks and 12 weeks of treatment

Secondary Objective :

* To evaluate the clinical and biological safety of valproate compared to lithium.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion criteria at Screening :

* Patients with a history of at least one manic episode in the previous three years or before the age of 60 for patients older than 60 at screening, as documented by medical records, or by a relative's report of information corroborating evidence of manic symptomatology for patients already known as bipolar patients. Newly diagnosed patients for bipolar disorder are allowed provided that the diagnosis is based on DSM IV TR[Diagnostic and Statistical Manual of Mental Disorders (DSM) fourth edition (IV)Text Revision (TR)]and that the patient is less than 30 years old.
* Patients with a current diagnosis of Bipolar I Disorder according to DSM IV TR
* Patients suffering from a current manic episode or a mixed episode according to DSM IV TR
* Patients with a minimum total score on the Young Mania Rating Scale (YMRS)of 18 at Screening

Inclusion criteria on D0 (Day 0):

* Patients having completed the wash-out period of at least 1 day duration (except for patients receiving no psychiatric treatment or a benzodiazepine at a dose lower than the equivalence of 8 mg of lorazepam and except for patients who only received injectable long-acting neuroleptics at least 7 days prior to Screening)
* Patients with a minimum total score on the Young Mania Rating Scale (YMRS) of 18 at D0

Exclusion criteria at Screening :

* Participation in a clinical trial within the three previous months
* Patients with a history of valproate intolerance defined as valproate discontinuation due to medically significant adverse effects
* Patients with a history of lithium intolerance defined as lithium discontinuation due to medically significant adverse effects
* Patients with a Central Nervous System (CNS) neoplasm, demyelinating disease, degenerative neurological disorder, active CNS infection or any progressive disorder that may blur interpretation of the study results
* Patients with a history of seizure disorder, cerebrovascular disease, structural brain damage from trauma, clinically significant focal neurological abnormalities, known EEG (Electroencephalography) with frank paroxysmal activity or a known CT scan of the brain demonstrating gross structural abnormalities
* Patients with uncontrolled gastro-intestinal, renal, hepatic, endocrine, cardiovascular, pulmonary, immunological or hematological disease
* Patients with renal insufficiency, cardiac insufficiency and Addison's disease
* Patients with past or current pancreatitis
* Patients with acute hepatitis, chronic hepatitis, or family history of severe hepatitis especially drug related, hepatic porphyry
* Patients with a current DSM IV diagnosis of alcohol or substance dependence (with the exception of nicotine or caffeine dependence) or substance abuse with stimulants including but not limited to cocaine, heroin, crack, amphetamines, pseudo-ephedrine, cold medications with phenylephrine or other stimulants. Alcohol or marijuana abuse prior to study entry will be accepted if related to the current manic episode, based on the investigator's judgment
* Pregnancy or lactation. Women of child bearing age should therefore be using a reliable contraceptive method
* Patients that require more than 300 mg of aspirin per day
* Patients with a medical condition which requires the continuous use of a treatment which could interfere with the safety or efficacy evaluation of valproate (anticonvulsant or anticoagulant therapy, zidovudine) or lithium (angiotensin converting enzyme inhibitors, tetracycline, reserpine, calcium channel blockers, triptans)
* Patients who received injectable long-acting neuroleptics less than 7 days prior to Screening
* Patients necessitating an Electro Convulsive Therapy
* Congenital prolongation of the QT interval

Exclusion criteria on D0 :

* Patients treated with an antidepressant within 5 days prior to randomization (D0)or with fluoxetine within 20 days preceding D0
* Patients with alterations of laboratory tests of potential significance:

  * ASAT or ALAT > 3 ULN (Upper Limit of Normal)
  * Alkaline phosphatase level > 1.5 ULN
  * Serum creatinine > or = to 150 µmol/l
  * Hemoglobin < 12 g/dl (men) and <11 g/dl (women)
  * Platelets < 150 000 /mm3
  * Neutrophils < 1 500 /mm3
  * Prothrombin time < 75 %
  * TSH (Thyroid-Stimulating Hormone)out of normal ranges
* QTc Bazett > 450 ms for male and > 470 ms for female on ECG (Electrocardiogram).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2004-02; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to D END in the Young Mania Rating Scale total score

SECONDARY OUTCOMES:
Change from baseline to each assessment in the YMRS score
Percentage of responders defined by a decrease of at least 50% in the YMRS score between D0 and D END
Percentage of responders at week 3 defined by a decrease of at least 50 % in the YMRS score between D0 and D21
Change in the Clinical Global Impressions Scale for Bipolar Disorder (CGI-BP) (20) between D0 and D21
Change in the CGI-BP between D0 and D END
Change in the MADRS between D0 and D21 (MADRS: Montgomery and Asberg Depression Rating Scale )
Change in the MADRS between D0 and D END
Survival analyses: Time to achieve 50% and 30% improvement in the YMRS score; Time to antidepressant intake; Time to drop-out for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Robert MANFREDI, MD, Study Director — Sanofi